CLINICAL TRIAL: NCT06506149
Title: A Prospective Evaluation of Microwave Ablation (MWA) in the Treatment of Relapsed Graves' Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Man Him Matrix Fung, Clinical Assistant Professor, The University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UW 23-343
Record Dates: First submitted 2024-07-11; First posted 2024-07-17 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-07

CONDITIONS: Graves Disease; Minimally Invasive Treatment; Ablation Treatment
Keywords: Graves disease; Thyroid function; remission; non surgical
MeSH Terms: conditions — Graves Disease

STUDY DESIGN:
Intervention Model Description: Consecutive patients with relapsed Graves' disease will be considered for microwave ablation treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Microwave ablation treatment (Experimental): All participants will be treated by a device for USG-guided Microwave ablation treatment
  Interventions: Device: Microwave ablation(MWA) device

INTERVENTIONS:
Device: Microwave ablation(MWA) device — The device for USG-guided MWA treatment would be performed under USG guidance, aiming to ablate the entire thyroid gland, i.e. the right lobe, left lobe, isthmus and pyramidal lobe.

SUMMARY:
Graves' disease is the most common cause of hyperthyroidism, with conventional treatment options being anti-thyroid drugs (ATD), radioiodine (RAI) and surgery. For ATD, it has been the first-line treatment over decades. Despite its ability to induce remission, minor side effects such as skin rash, gastrointestinal disturbance and arthralgia occur in around 5% of patients, while serious adverse reactions including agranulocytosis and hepatotoxicity are potentially life threatening. Patients are usually treated with ATD for 12 to 18 months but the relapse rate was reported to be up to 50-60% which these patients would require more definitive treatment options with RAI or thyroidectomy. However, RAI is not preferable in patients with Graves' ophthalmopathy as it could further worsen eye symptoms. RAI may also cause hypothyroidism in a substantial proportion of patients, with a subsequent need for lifelong thyroxine replacement. As for thyroidectomy, it carries an overall 2-10% risk of complications including bleeding, transient or permanent recurrent laryngeal nerve injury and hypoparathyroidism. Due to the drawbacks of the various conventional treatment options, there has been increasing interest in the development of minimally invasive treatment alternatives in recent years. With the evolution of thermal ablative strategies, high-intensity focused ultrasound (HIFU) and radiofrequency ablation (RFA) have been reported as feasible treatment options for relapsed Graves' disease. There has also been increasing reports in the use of microwave ablation (MWA) in the treatment of benign thyroid nodules. MWA works via generation of electromagnetic field and is performed by inserting a microwave antenna into the thyroid gland percutaneously under ultrasound (USG) guidance. The active tip of the antenna causes oscillation of the surrounding water molecules which induces frictional heat and creates a thermal ablative effect. As compared to RFA, MWA is not affected by heat sink effect and may require a shorter treatment time. Similar to other thermal ablative approaches, MWA has the merits of avoiding surgical scar, organ preservation as well as being an ambulatory procedure.

ELIGIBILITY:
Inclusion Criteria:

* (a) age older than 18 years,
* (b) relapsed Graves' disease despite an adequate ATD treatment for 18 months or more
* (c) absence of vocal cord immobility

Exclusion Criteria:

* (a) patients who prefer or are indicated for surgery,
* (b) presence of head and/or neck disease preventing hyperextension of the neck,
* (c) history of thyroid cancer or other malignant tumours in the neck region,
* (d) history of neck irradiation,
* (e) severe Graves' ophthalmopathy,
* (f) large compressive goitre,
* (g) pregnancy or lactation, and
* (h) any contraindication to intravenous sedation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2023-07-04 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
To measure the remission rate of Graves' disease at 6-months post-procedure | 6 months
  To measure the remission rate of Graves' disease at 6-months post-procedure

SECONDARY OUTCOMES:
Change of quality of life by SF12 ver 2 | 6 months
  SF-12(v2) is an assessment tool about quality of life. It comprises 12 question items ranging from 11 (worst quality of life) to 56 (best quality of life).
To measure the percentage of volume change | 6 months
  the percentage of volume change would be calculated as: ([Volbasal - Volfinal] · 100)/Volbasal.

CONTACTS AND LOCATIONS:
Locations (1):
- Queen Mary Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Anticipate from June 30, 2026 for 1 years at least

REFERENCES:
- [Background] Cooper DS. Antithyroid drugs. N Engl J Med. 2005 Mar 3;352(9):905-17. doi: 10.1056/NEJMra042972. No abstract available. PMID 15745981
- [Background] Yip J, Lang BH, Lo CY. Changing trend in surgical indication and management for Graves' disease. Am J Surg. 2012 Feb;203(2):162-7. doi: 10.1016/j.amjsurg.2011.01.029. Epub 2011 Jun 17. PMID 21683939
- [Background] Lang BH, Woo YC, Chiu KW. Two-year outcomes of single-session high-intensity focused ultrasound (HIFU) treatment in persistent or relapsed Graves' disease. Eur Radiol. 2019 Dec;29(12):6690-6698. doi: 10.1007/s00330-019-06303-8. Epub 2019 Jun 17. PMID 31209622
- [Background] Lang BH, Woo YC, Wong IY, Chiu KW. Single-Session High-Intensity Focused Ultrasound Treatment for Persistent or Relapsed Graves Disease: Preliminary Experience in a Prospective Study. Radiology. 2017 Dec;285(3):1011-1022. doi: 10.1148/radiol.2017162776. Epub 2017 Jul 20. PMID 28727542
- [Background] Fung MHM, Lang BHH. Efficacy of single-session radiofrequency ablation (RFA) in rendering euthyroidism for persistent/relapsed Graves' disease, a pilot study. Eur Radiol. 2023 Sep;33(9):6534-6544. doi: 10.1007/s00330-023-09620-1. Epub 2023 Apr 10. PMID 37036479
- [Background] Orloff LA, Noel JE, Stack BC Jr, Russell MD, Angelos P, Baek JH, Brumund KT, Chiang FY, Cunnane MB, Davies L, Frasoldati A, Feng AY, Hegedus L, Iwata AJ, Kandil E, Kuo J, Lombardi C, Lupo M, Maia AL, McIver B, Na DG, Novizio R, Papini E, Patel KN, Rangel L, Russell JO, Shin J, Shindo M, Shonka DC Jr, Karcioglu AS, Sinclair C, Singer M, Spiezia S, Steck JH, Steward D, Tae K, Tolley N, Valcavi R, Tufano RP, Tuttle RM, Volpi E, Wu CW, Abdelhamid Ahmed AH, Randolph GW. Radiofrequency ablation and related ultrasound-guided ablation technologies for treatment of benign and malignant thyroid disease: An international multidisciplinary consensus statement of the American Head and Neck Society Endocrine Surgery Section with the Asia Pacific Society of Thyroid Surgery, Associazione Medici Endocrinologi, British Association of Endocrine and Thyroid Surgeons, European Thyroid Association, Italian Society of Endocrine Surgery Units, Korean Society of Thyroid Radiology, Latin American Thyroid Society, and Thyroid Nodules Therapies Association. Head Neck. 2022 Mar;44(3):633-660. doi: 10.1002/hed.26960. Epub 2021 Dec 23. PMID 34939714
- [Background] Song YN, Shi WY, Chen JJ, Wang Q, Li XQ, Liu M, Cao BY, Ni X, Gong CX. [A case of ultrasound-guided microwave ablation for Graves disease]. Zhonghua Er Ke Za Zhi. 2022 Oct 2;60(10):1081-1082. doi: 10.3760/cma.j.cn112140-20220301-00166. Chinese. PMID 36207860
- [Background] Zhu JE, Zhang HL, Yu SY, Xu HX. US-guided percutaneous microwave ablation for hyperthyroidism and immediate treatment response evaluation with contrast-enhanced ultrasound. Clin Hemorheol Microcirc. 2021;79(3):435-444. doi: 10.3233/CH-211180. PMID 34092625
- [Background] Dighe M, Barr R, Bojunga J, Cantisani V, Chammas MC, Cosgrove D, Cui XW, Dong Y, Fenner F, Radzina M, Vinayak S, Xu JM, Dietrich CF. Thyroid Ultrasound: State of the Art Part 1 - Thyroid Ultrasound reporting and Diffuse Thyroid Diseases. Med Ultrason. 2017 Jan 31;19(1):79-93. doi: 10.11152/mu-980. PMID 28180201
- [Background] Du JR, Li WH, Quan CH, Wang H, Teng DK. Long-term outcome of microwave ablation for benign thyroid nodules: Over 48-month follow-up study. Front Endocrinol (Lausanne). 2022 Aug 1;13:941137. doi: 10.3389/fendo.2022.941137. eCollection 2022. PMID 35979439
- [Background] Zhao J, Qian L, Liu Y, Tan X. A long-term retrospective study of ultrasound-guided microwave ablation of thyroid benign solid nodules. Int J Hyperthermia. 2021;38(1):1566-1570. doi: 10.1080/02656736.2021.1994659. PMID 34727816